CLINICAL TRIAL: NCT04728672
Title: The Effects of Kinesio Taping on Hip Abductor Muscle Strength and EMG Activity in Athletes With Chronic Ankle Instability
Brief Title: Effects of Kinesio Taping on Hip Abductor Muscle Strength and EMG Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Masood Khan, Principal Investigator, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RRC-2019-27
Record Dates: First submitted 2021-01-24; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Chronic Ankle Instability
Keywords: Chronic ankle instability; Hip abductors; Kinesio Taping; Muscle strength; EMG
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Intervention Model Description: Two parallel groups pretest-posttest design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Kinesio tape was applied and then outcome measures were noted.
  Interventions: Other: Kinesio Tape
- Control Group (Placebo Comparator): Placebo Micropore Tape was applied and then outcome measures were noted.
  Interventions: Other: Micropore Tape

INTERVENTIONS:
Other: Kinesio Tape — Kinesio Tape
  Arms: Experimental Group
Other: Micropore Tape — Micropore Tape
  Arms: Control Group

SUMMARY:
Athletes with chronic ankle instability tend to develop Glutei muscle weakness. This weakness makes the lower limb prone to injuries. Kinesio Tape (KT) may assist this muscle in performing its functions thus preventing injuries.

DETAILED DESCRIPTION:
The aim was to study the effects of Kinesio Tape on hip abductor muscle strength and EMG activity. Pretest-posttest experimental design was used. The study was conducted in the research lab of the University. Thirty-four athletes with a mean age of 22.08 years participated in the study. For the experimental group Kinesio Tape and for the control group Micropore Tape (MT) was applied over Gluteus Medius (GM) muscle. GM muscle's strength and EMG activity were noted in supine and during the Single-Leg Squat Test (SLST) respectively before and after the intervention. Hip abductor muscle strength measured through a maximum voluntary isometric contraction (MVIC) and GM activation measured through EMG. Handheld dynamometer (Lafayette manual muscle test system), Power Lab EMG system.

ELIGIBILITY:
Inclusion Criteria:

* Repeated episodes of giving way after an initial ankle sprain,
* A history of at least 2 ankle sprains to the same side without injury to the contralateral ankle in the last 2 years,
* No history of other trauma to the lower extremities for the past 3 months prior to the study,
* Participants also needed to be capable of full weight-bearing without analgia,
* Subjectively reported that functional use of ankle had plateaued since the last injury.

Exclusion Criteria:

* Participants having a history of ankle fracture, knee ligament injury, back or lower limb surgery, neuromuscular disease, or current neurological deficit,
* Currently receiving ankle rehabilitation were excluded from the study.

Ages: 18 Years to 26 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-12 (Actual); Primary Completion 2020-11-23 (Actual); Study Completion 2020-12-17 (Actual)

PRIMARY OUTCOMES:
Maximum Voluntary Isometric Contraction | upto 1 month
  Participants exerted maximum resistance against the dynamometer in the direction of hip abduction
Electromyography | upto 1 month
  Electromyographic activity of gluteus medius was measured during single leg squat test

CONTACTS AND LOCATIONS:
Overall Officials: Masood Khan, MPTh, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No